CLINICAL TRIAL: NCT04606927
Title: Pragmatic Urinary Sodium-based Treatment algoritHm in Acute Heart Failure
Acronym: PUSH-AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jozine ter Maaten, Principle investigator, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020000710
Record Dates: First submitted 2020-10-18; First posted 2020-10-28 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure Acute
Keywords: loop diuretics; natriuresis
MeSH Terms: interventions — Natriuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natriuresis guided treatment (Active Comparator)
  Interventions: Other: Natriuresis
- Standard of care (No Intervention)

INTERVENTIONS:
Other: Natriuresis — Patients with insufficient decongestive response based on natriuresis (in the active arm) will be eligible for treatment adjustments according to the natriuresis guided treatment algorithm.
  Arms: Natriuresis guided treatment

SUMMARY:
Administration of loop diuretics to achieve decongestion is the current cornerstone of therapy for acute heart failure. Unfortunately, there is a lack of evidence of how to guide diuretic treatment. Recently, urinary sodium, as a response measure of diuretic response, has been proposed as a target for therapy. The hypothesis of this study is that natriuresis guided therapy in patients with acute heart failure will improve diuretic response, decongestion, and reduce length of hospital stay, as well as heart failure rehospitalisations.

DETAILED DESCRIPTION:
Objective: To assess the effect of natriuresis guided therapy in acute heart failure to improve diuretic response, decongestion, and clinical outcomes

Study design: Randomised, controlled, open label study

Study population: 310 patients admitted with the primary diagnosis of acute heart failure requiring intravenous loop diuretics.

Intervention: natriuresis guided treatment versus standard of care

Main study parameters/endpoints:

Co-primary outcome: total natriuresis after 24 hours, and first occurrence of all-cause mortality or heart failure rehospitalisation at 6 months Secondary outcomes: 48- and 72-hours natriuresis, length of hospital stay, percentage change in NT-proBNP at 48 and 72 hours.

Safety endpoint: doubling of serum creatinine at 24 or 48 hours, worsening heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Primary diagnosis of acute /decompensated heart failure as assessed by treating physician

   a. Acute Heart failure can be de novo or exacerbation of known heart failure and diagnosis is based on criteria in the ESC HF guidelines
3. Requirement of intravenous diuretic use

Exclusion Criteria:

1. Dyspnoea primarily due to non-cardiac causes
2. Patients with severe renal impairment receiving dialysis or requiring ultrafiltration
3. Inability to follow instructions
4. Any other medical conditions that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ter Maaten JM, Beldhuis IE, van der Meer P, Krikken JA, Postmus D, Coster JE, Nieuwland W, van Veldhuisen DJ, Voors AA, Damman K. Natriuresis-guided diuretic therapy in acute heart failure: a pragmatic randomized trial. Nat Med. 2023 Oct;29(10):2625-2632. doi: 10.1038/s41591-023-02532-z. Epub 2023 Aug 28. PMID 37640861

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of care
Period: Overall Study
Arm/Group | Natriuresis Guided Treatment | Standard of Care
Started | 150 | 160
Completed | 150 | 160
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natriuresis Guided Treatment | Standard of Care | Total
Number analyzed (Participants) | 150 | 160 | 310
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [66 to 82] | 74 [65 to 81] | 74 [65 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 77 | 138
  Male | 89 | 83 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 142 | 155 | 297
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Netherlands | 150 | 160 | 310

OUTCOME MEASURES:

1. Primary Outcome: Total Natriuresis After 24 Hours
Description: The first component of the co-primary end-point is total natriuresis after 24 h (mmol). To assess this, urine is collected for 24 hours after the first administration of diuretics according to the study protocol and natriuresis is calculated as the total amount of diuresis (L) multiplied by the urinary sodium concentration (mmol/L).
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Natriuresis Guided Treatment | Standard of Care
Number analyzed (Participants) | 131 | 147
mmol | 409 (178) | 345 (202)

2. Primary Outcome: First Occurrence of All-cause Mortality or Heart Failure Rehospitalization After 180 Days
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Natriuresis Guided Treatment | Standard of Care
Number analyzed (Participants) | 150 | 159
Participants | 46 | 50

3. Secondary Outcome: 48-hours Natriuresis
Description: 48-hour natriuresis will be assessed by collecting urine for a second period of 24 hours after the first 24-hour urine collection according to the study protocol and natriuresis is calculated as the total amount of diuresis (L) multiplied by the urinary sodium concentration (mmol/L).
Time Frame: 48 hours
Reporting Status: Not Posted

4. Secondary Outcome: 72-hours Natriuresis
Description: 72-hour natriuresis will be assessed by collecting urine for a third period of 24 hours after the second 24-hour urine collection according to the study protocol and natriuresis is calculated as the total amount of diuresis (L) multiplied by the urinary sodium concentration (mmol/L).
Time Frame: 72 hours
Reporting Status: Not Posted

5. Secondary Outcome: Length of Hospital Stay
Description: Number of days of the index hospitalization
Time Frame: Variable
Reporting Status: Not Posted

6. Secondary Outcome: Percentage Change in NT-proBNP at 48 Hours
Description: Relative NT-proBNP change (%) after 48 hours compared with baseline
Time Frame: 48 hours
Reporting Status: Not Posted

7. Secondary Outcome: Percentage Change in NT-proBNP at 72 Hours
Description: Relative NT-proBNP change (%) after 72 hours compared with baseline
Time Frame: 72 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Safety Endpoint: Doubling of Serum Creatinine at 24 Hours
Description: The first safety endpoint is defined as number of patients with a doubling of serum creatinine at 24 hours compared with baseline serum creatinine.
Time Frame: 24 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Safety Endpoint: Doubling of Serum Creatinine at 48 Hours
Description: The second safety endpoint is defined as the number of patients with a doubling of serum creatinine at 48 hours compared with baseline serum creatinine.
Time Frame: 48 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Worsening Heart Failure
Description: The third safety endpoint is defined as the number of patients with worsening heart failure during hospitalization.
Time Frame: During the index hospitalization (variable)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the study period (6 months)
Arm/Group | Natriuresis Guided Treatment | Standard of Care
All-Cause Mortality (participants affected / at risk) | 29/150 | 33/160
Serious Adverse Events (participants affected / at risk) | 60/150 | 70/160
Other Adverse Events (participants affected / at risk) | 0/150 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natriuresis Guided Treatment (N=150) | Standard of Care (N=160)
Diverse (Cardiac disorders) | 60 (60) | 70 (70)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natriuresis Guided Treatment (N=150) | Standard of Care (N=160)
Other (Cardiac disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT04606927/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT04606927/SAP_001.pdf